CLINICAL TRIAL: NCT04113278
Title: Role of Fibirnogen Like Protein 2 as Aprognostic Factor in High Grade Glioma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: sohaila Essam (Other)
Responsible Party: Sponsor-Investigator, sohaila Essam, Role of fibrinogen like protein 2 as aprognostic factor in high grade glioma, Assiut University
Organization: Assiut University (Other)
Other Study IDs: FGL2 in brain cancer
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Brain Tumor Adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: FGL2 immunohisyochemistry — Correlation between FLG2 expression and progression free survival and overall surviv

SUMMARY:
The study population was selected from high grade glioma pateints attending the Department of Clinical Oncology, Assiut University hospital during the period from December 2018 to September 2020, we analyzed human high grade gliomas paraffin block for FLG2 expression

DETAILED DESCRIPTION:
Glioblastoma is the most common malignant primary brain tumor in adults, and despite aggressive treatment, it is incurable Patient prognosis differs considerably within the different World Health Organization (WHO) grades, poorest prognosis for patients with the grade IV tumour- the glioblastoma multiform (GBM).

Fibrinogen-like protein 2 (FGL2),regulates both innate and adaptive immunity. FGL2 is a 439 amino acid secreted protein that is similar to the β- and γ-chains of fibrinogen.

Secreted FGL2 (sFGL2) is the key regulator in immunosuppression may play important role in malignant transformation of low to high by inhibiting the proliferation of T cell Study the role of fibrinogen-like protein2 on Immunosuppression and progression ，free survival and overall survival in high grade glioma

ELIGIBILITY:
Inclusion Criteria:

* Pateints>18 years old
* Pathologically proven high grade glioma
* Total or subtotal resection of the tumor
* Patients received concurrent radiation therapy with temozolomide followed by adjuvant temozolamide for 6 months

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Other comorbidity
* Previous malignancy or radiation therapy or chemotherapy

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population was selected from high grade glioma pateints attending the Department of Clinical Oncology, Assiut University hospital during the period from December 2018 to September 2020, we analyzed human high grade gliomas paraffin block for FLG2 expression
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Rple of FGL2in high grade glioma as aprognostic factor | baseline
  Correlation between FLG2 expression and progression free survival and overall survival

REFERENCES:
- [Background] Latha K, Yan J, Yang Y, Gressot LV, Kong LY, Manyam G, Ezhilarasan R, Wang Q, Sulman EP, Eric Davis R, Huang S, Fuller GN, Rao A, Heimberger AB, Li S, Rao G. The Role of Fibrinogen-Like Protein 2 on Immunosuppression and Malignant Progression in Glioma. J Natl Cancer Inst. 2019 Mar 1;111(3):292-300. doi: 10.1093/jnci/djy107. PMID 29947810
- [Background] Yan J, Zhao Q, Gabrusiewicz K, Kong LY, Xia X, Wang J, Ott M, Xu J, Davis RE, Huo L, Rao G, Sun SC, Watowich SS, Heimberger AB, Li S. FGL2 promotes tumor progression in the CNS by suppressing CD103+ dendritic cell differentiation. Nat Commun. 2019 Jan 25;10(1):448. doi: 10.1038/s41467-018-08271-x. PMID 30683885